CLINICAL TRIAL: NCT05504603
Title: A Phase 2 Study of Zanubrutinib-rituximab(ZR) in Patients With Newly Diagnosed Untreated Mantle Cell Lymphoma
Brief Title: Zanubrutinib-rituximab(ZR) in Patients With Newly Diagnosed Untreated Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jinzm 004
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Untreated Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Zanubrutinib; Rituximab; ASCT
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zanubrutinib(80mg), rituximab(100mg), ASCT (Experimental): 1. Phase I(Combined Immunotherapy Phase):
     Part A(Induction Immunotherapy Phase): Patients receive zanubrutinib on days 1-28 and rituximab on day 1,8,15,22.
     Part B(Consolidation Immunotherapy Phase): Patients receive zanubrutinib on days 1-28 and rituximab on day 1. Treatment cycles repeat every 28 days for 4 cycles.
  2. Phase II(ASCT): BEAM pretreatment. Patients receive semustine on day1, etoposide on days 2-5, cytarabine on days 2-5 and melphalan on day 6.
  3. Phase III(maintenance): Zanubrutinib
  Interventions: Drug: zanubrutinib and rituximab; Drug: BEAM pretreatment; Drug: zanubrutinib maintenance

INTERVENTIONS:
Drug: zanubrutinib and rituximab — zanubrutinib 160mg PO BID d1-28; rituximab 375mg/m2 IVGTT d1,8,15,22. Other name: Part A
Drug: zanubrutinib and rituximab — zanubrutinib 160mg PO BID d1-28; rituximab 375mg/m2 IVGTT d1. Other name: Part B
Drug: BEAM pretreatment — semustine 250mg/m2 PO d1; etoposide 200mg/m2 IV d2-5; cytarabine 400mg/m2 IV d2-5; melphalan 140mg/m2 IV d6.
Drug: zanubrutinib maintenance — zanubrutinib 160mg PO BID.

SUMMARY:
The proposed study is a prospective, single-center, single-arm and open-ended phase II study in patients over the age of 18 with previously untreated mantle cell lymphoma(MCL). The primary objective of this study is to explore the safety and efficacy of a new chemo-free treatment pattern zanubrutinib-rituximab(ZR) in newly diagnosed MCL.

DETAILED DESCRIPTION:
The study will start with an initial 28-days of induction immunotherapy with ZR and 4 cycles of consolidation immunotherapy with ZR，following imaging examinations to evaluate response rates. Patients who are evaluated as SD and PD will be withdrawn from the trial,while those who achieve PR and CR will be further stratified according to their age and physical status. The older or frail patients who are ineligible for ASCT will take zanubrutinib orally until intolerable toxicity or disease progression. Patients who are young and fit for transplantation will receive ASCT consolidation. After ASCT, patients with CR will end therapy and enter the follow-up stage, while patients with PR will continue to take zanubrutinib orally until intolerable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or Cytologically confirmed Mantle Cell Lymphoma(excluding indolent Mantle Cell Lymphoma) by the 2008 World Health Organization (WHO) Classification of diseases;
2. Initial untreated patients;
3. Age ≥ 18 years;
4. ECOG score 0-2;
5. Women must not be pregnant or breastfeeding and agree to avoid pregnancy prior to study entry, for the duration of study participation, and for 12 months thereafter. Male patients must agree that their spouses will not become pregnant during the study period and for 12 months thereafter;
6. Patients must have measurable disease (i.e., ≥ 1.0 cm in lymph nodes diameter; or skin lesions assessed by physical examination);
7. Written informed consent obtained from the subject.

Exclusion Criteria:

1. Indolent Mantle Cell Lymphoma;
2. Patients with severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine > 3 times the upper limit of normal)
3. Uncontrolled active infection, with the exception of tumor-related B symptom fever;
4. Patients with organic heart disease with clinical symptoms or cardiac dysfunction (NYHA grade ≥2);
5. Co-existence of other tumors;
6. Any other psychological conditions that prevent patients from participating in the study or signing the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-07-26 (Estimated); Study Completion 2025-07-26 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) in all patients | At the end of cycle 3 and cycle 5(each cycle is 28 days)
  The rate of patients who achieved complete response and partial response after ZR combined immunotherapy
Complete Response Rate(CRR) in all patients | At the end of cycle 3 and cycle 5(each cycle is 28 days)
  The rate of patients who achieved complete response after ZR combined immunotherapy.
Overall Response Rate(ORR) in patients received ASCT | 1 month after ASCT
  The rate of patients who achieved complete response and partial response after ASCT.
Complete Response Rate(CRR) in patients received ASCT | 1 month after ASCT
  The rate of patients who achieved complete response after ASCT.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months after the last patient's enrollment.
  OS will be assessed from the first ZR given to date of death or end of follow-up.
Progression Free Survival (PFS) | up to 24 months after the last patient's enrollment.
  PFS will be assessed from the first ZR given to date of progression, relapse, death or end of follow-up.
Incidence of Treatment-Emergent Adverse Events, Treatment-Related Adverse Events and Serious Adverse Events | initiation of study drug until 30 days after last dose.
  The safety and tolerability of the therapeutic regimen measured by the incidence of Treatment-Emergent Adverse Events, Treatment-Related Adverse Events and Serious Adverse Events.
Minimal Residual Disease (MRD) | At the end of cycle 5 ZR (each cycle is 28 days) and 1 month after ASCT.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available at the First Affiliated Hospital and other researchers after the end of the study.
Supporting Information: Study Protocol, SAP
Time Frame: after the end of the study